CLINICAL TRIAL: NCT02880865
Title: Immunogenicity and Safety of Concurrent Administration of Live, Attenuated SA 14-14-2 Japanese Encephalitis Vaccine and Measles-Mumps-Rubella Vaccine in Infants 9-12 Months of Age in the Philippines
Brief Title: Immunogenicity and Safety of Japanese Encephalitis Vaccine When Given With Measles-Mumps-Rubella (MMR) Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Research Institute for Tropical Medicine (Other Government); Syneos Health (Other); DFNet Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEV06; PHRR160822-001339 (Registry Identifier: Philippine Health Research Registry (PHRR))
Record Dates: First submitted 2016-08-17; First posted 2016-08-26 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-03

CONDITIONS: Encephalitis, Japanese; Measles; Mumps; Rubella
Keywords: vaccine
MeSH Terms: conditions — Encephalitis, Japanese; Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - MMR and CD-JEV (Experimental): Participants receiving one dose of CD-JEV vaccine and one dose of MMR vaccine concurrently at Day 0; Group 1 will also receive a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
  Interventions: Biological: Live attenuated SA 14-14-2 Japanese Encephalitis vaccine; Biological: Measles, mumps, rubella vaccine
- Group 2 - MMR then CD-JEV (Experimental): Participants receiving one dose of MMR vaccine at Day 0 and one dose of CD-JEV 56 days later. Group 2 will receive a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
  Interventions: Biological: Live attenuated SA 14-14-2 Japanese Encephalitis vaccine; Biological: Measles, mumps, rubella vaccine

INTERVENTIONS:
Biological: Live attenuated SA 14-14-2 Japanese Encephalitis vaccine — Single 0.5 mL dose of World Health Organization prequalified live, attenuated SA 14-14-2 JE vaccine manufactured by Chengdu Institute of Biological Products, Chengdu, China, administered by subcutaneous injection
  Other Names: CD-JEV; CD.JEVAX®; RS.JEV®
Biological: Measles, mumps, rubella vaccine — Single 0.5 mL dose of live, attenuated measles-mumps-rubella vaccine (Schwarz measles virus, RIT 4385 mumps strain, and Wistar RA 27/3 rubella virus) manufactured by GlaxoSmithKline, Inc., administered by subcutaneous injection.
  Other Names: MMR; Priorix®

SUMMARY:
This study aims to provide evidence that co-administration of measles-mumps-rubella vaccine (MMR) and live attenuated SA 14-14-2 Japanese encephalitis vaccine (CD-JEV) does not adversely affect immunogenicity or safety.

DETAILED DESCRIPTION:
When incorporating a new vaccine in the Expanded Programme on Immunization (EPI), it is important to provide evidence that it can be introduced concurrently with other routine pediatric vaccines without significantly impairing the immune response to any vaccine while maximizing coverage and minimizing cost. This non-inferiority study aims to compare CD-JEV and MMR responses in a population of children in a country where MMR introduction is ongoing or planned. This information will help the ministries of health evaluate the addition of CD-JEV into routine EPI.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 months to < 10 months at the time of enrollment.
* Residence in the study area.
* At least one parent or guardian willing to provide written informed consent.
* Generally healthy and free of obvious health problems as established by medical history, physical examination, and clinical judgment.
* A parent or guardian is willing to attend all planned study visits and allow home visits and phone contacts, as required by the protocol.

Exclusion Criteria:

* Previous receipt of any measles-mumps-rubella containing vaccine.
* Previous receipt of any Japanese encephalitis vaccine.
* History of measles, mumps, rubella, or Japanese encephalitis infection.
* Administration of any other vaccine within 28 days prior to administration of a study vaccine or planned vaccination of any vaccine other than catch-up doses of routine EPI vaccines or oral polio vaccine during the 28 days after study vaccination.
* History of allergic disease or known hypersensitivity to any component of the study vaccines and/or following administration of vaccines included in the local program of immunization.
* Use of any investigational or non-registered drug within 90 days prior to the administration of study vaccines or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within 90 days prior to the administration of study vaccines or planned administration during the study period.
* Chronic administration (defined as > 7 days) of immunosuppressing or other immune-modifying agents within 14 days before or after vaccination (including systemic corticosteroids equivalent to prednisone ≥ 0.5 mg/kg/day; topical and inhaled steroids are allowed).
* Primary or acquired immunodeficiency, including human immunodeficiency virus (HIV) infection, or a family history of congenital or hereditary immunodeficiency as reported by parent.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history or physical examination, which might interfere with the study objectives.
* Severely malnourished infants as measured by World Health Organization weight-for-height tables (Z-score < -3).
* Any condition or criterion that, in the opinion of the study physician, might compromise the well-being of the participant, compliance with study procedures, or interpretation of the outcomes of the study.
* Acute illness at the time of enrollment defined as the presence of a moderate or severe illness with fever (axillary temperature ≥ 38.0°C) or without fever (severity determined at the discretion of the study physician). Acute illness is a temporary exclusion. Vaccination should be postponed at least 7 days after recovery. A visit for reassessment may be scheduled 7 days or more after temporary exclusion illness is resolved. Eligibility for study participation must be reassessed again at the next visit.

Ages: 9 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 628 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Capeding, MD, Principal Investigator — Research Institute for Tropical Medicine
Locations (1):
- Research Institute for Tropical Medicine, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No
The study team agrees that the practice of offering study results to participants in human research is fundamental to the ethical principle of respect for persons. However, the sponsor prefers to report at the aggregate level to maintain participant confidentiality and ensure results are community-based. Thus, the sponsor plans to report results at the aggregate level. The sponsor will produce a poster of the results to be placed at each health center. A community meeting may also be held to communicate the results. Aggregate results will also be posted on www.clinicaltrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 health centers in the Philippines.
Pre-assignment Details: Filipino children aged 9 to < 10 months were randomized in a 1:1 ratio to receive measles, mumps, and rubella vaccine (MMR) and prequalified live, attenuated SA-14-4-2 Japanese encephalitis vaccine (CD-JEV) together (Group 1) or 56 days apart (Group 2). All participants received a second dose of MMR at 12 months of age.
Groups:
- Group 1: MMR and CD-JEV: Participants received one dose of CD-JEV vaccine and one dose of MMR vaccine concurrently at Day 0. Participants received a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
- Group 2: MMR Then CD-JEV: Participants received one dose of MMR vaccine at Day 0 and one dose of CD-JEV 56 days later. Participants received a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
Period: Overall Study
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Started | 314 | 314
Received MMR Dose 1 | 314 | 314
Received CD-JEV | 314 | 309
Received MMR Dose 2 | 313 | 311
Completed | 313 | 311
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV | Total
Number analyzed (Participants) | 314 | 314 | 628
Age, Continuous [Median (Full Range); unit: months] | 9.2 [9.0 to 10.0] | 9.2 [9.0 to 10.0] | 9.2 [9.0 to 10.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 157 | 301
  Male | 170 | 157 | 327
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Philippines | 314 | 314 | 628

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Measles Seropositivity 56 Days Post-vaccination
Description: Measles immunogenicity was assessed by the percentage of participants with demonstrated seropositivity for measles at 56 days post-vaccination. Seropositivity was defined by a concentration of ≥ 120 mIU/mL of anti-measles neutralizing antibody titer, as measured by the plaque reduction neutralization test (PRNT) (dilution converted to concentration using the 3rd International Standard Reference serum).
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: The measles per-protocol population included participants who fulfilled the eligibility criteria, received all study vaccines as assigned, provided valid measles serology results at baseline and Day 56, did not take any prohibited concomitant medications within 28 days post-vaccination, and did not show measles seropositivity at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 311 | 306
percentage of participants | 98.1 [95.8 to 99.3] | 98.0 [95.8 to 99.3]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; The primary hypotheses evaluated the non-inferiority of the concomitant administration of MMR and CD-JEV vaccines (Group 1) to MMR and CD-JEV vaccines given 2 months apart (Group 2) in children 9 months of age at 56 days in terms of percentage of participants achieving seropositivity to measles and rubella assuming a non-inferiority margin of 10%; Test type: Non-Inferiority — Non-inferiority was achieved if the lower limit of the two-sided 95% confidence interval (CI) for the difference in percentages of participants with seropositivity between the two groups (concurrent administration minus separate administration) at 56 days post-vaccination was > -10% for both measles and rubella results; Difference = 0.0, 95% CI 2-sided [-2.1 to 2.2]

2. Primary Outcome: Percentage of Participants With Rubella Seropositivity 56 Days Post-vaccination
Description: Rubella immunogenicity was assessed by the percentage of participants with demonstrated seropositivity for rubella at 56 days post-vaccination. Seropositivity was defined as antirubella immunoglobulin G (IgG) concentration of ≥ 10 IU/mL (corresponding to an optical density ratio ≥ 1.10) using a commercial IgG enzyme-linked immunosorbent assay (ELISA).
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: The rubella per-protocol population included participants who fulfilled the eligibility criteria, received all study vaccines as assigned, provided valid rubella serology results at baseline and Day 56, did not take any prohibited concomitant medications within 28 days post-vaccination, and did not show rubella seropositivity at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 285 | 295
percentage of participants | 100.0 [98.7 to 100.0] | 99.7 [98.1 to 100.0]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority was achieved if the lower limit of the two-sided 95% CI for the difference in percentages of participants with seropositivity between the two groups (concurrent administration minus separate administration) at 56 days post-vaccination was > -10% for both measles and rubella results; Difference = 0.3, 95% CI 2-sided [-0.3 to 1.0]

3. Secondary Outcome: Percentage of Participants With Mumps Seropositivity 56 Days Post-vaccination
Description: Mumps immunogenicity was assessed by the percentage of participants with demonstrated seropositivity for mumps at 56 days post-vaccination. Seropositivity was defined as an optical density ratio ≥ 1.10 using a commercial ELISA.
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: The mumps per-protocol population included participants who fulfilled eligibility criteria, received all study vaccines as assigned, provided valid mumps serology results at baseline and Day 56, did not take any prohibited concomitant medications within within 28 days post-vaccination, and did not show mumps seropositivity at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 270 | 265
percentage of participants | 98.5 [96.3 to 99.6] | 98.5 [96.2 to 99.6]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Non-Inferiority — The percentage of participants with seropositivity for mumps at 56 days post-vaccination between Group 1 and Group 2 were compared using a non-inferiority test. Non-inferiority of Group 1 to Group 2 in terms of seropositivity for mumps was demonstrated if the lower limit of the two-sided 95% CI for the difference of seropositivity rates between the two groups (concurrent administration minus separate administration) at 56 days post-vaccination was > -10%; Difference = 0.0, 95% CI 2-sided [-2.0 to 2.1]

4. Secondary Outcome: Geometric Mean Concentration (GMC) for Anti-measles Neutralizing Antibody Concentration at 56 Days Post-vaccination
Description: Anti-measles neutralizing antibody concentration was measured by the plaque reduction neutralization test (PRNT).
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 311 | 306
mIU/mL | 1964.4 [1769.3 to 2181.0] | 1866.3 [1649.1 to 2112.0]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; GMC Ratio = 1.1, 95% CI 2-sided [0.9 to 1.2] — Group 1/Group 2 ratio obtained using analysis of covariance (ANCOVA) with log10-transformed antibody concentration as dependent variable and treatment group as the explanatory variable adjusted for log10-transformed baseline antibody concentration

5. Secondary Outcome: GMC for Anti-rubella IgG Antibody Concentration at 56 Days Post-vaccination
Description: Anti-rubella immunoglobulin G (IgG) concentration was measured using a commercial IgG enzyme-linked immunosorbent assay (ELISA).
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 285 | 295
IU/mL | 230.8 [214.4 to 248.5] | 229.8 [210.0 to 251.3]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; GMC Ratio = 1.0, 95% CI 2-sided [0.9 to 1.1] — Group 1/Group 2 ratio obtained using an ANCOVA method with log 10-transformed antibody concentration as dependent variable and treatment group as explanatory variable adjusted for log 10-transformed baseline antibody concentration

6. Secondary Outcome: Seroconversion Rate for Measles 56 Days Post-vaccination
Description: The seroconversion rate for measles at 56 days post-vaccination was defined as the percentage of participants with a change in serostatus from negative to positive 56 days after vaccination or a four-fold rise in concentration 56 days after vaccination if seropositive for measles at baseline. Seropositivity was defined by a concentration of ≥ 120 mIU/mL of anti-measles neutralizing antibody titer, as measured by the plaque reduction neutralization test (PRNT).
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 311 | 306
percentage of participants | 98.1 [95.8 to 99.3] | 98.0 [95.8 to 99.3]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; Difference = 0.0, 95% CI 2-sided [-2.1 to 2.2] — Group 1 - Group 2

7. Secondary Outcome: Seroconversion Rate for Mumps 56 Days Post-vaccination
Description: The seroconversion rate for mumps at 56 days post-vaccination was defined as the percentage of participants with a change in serostatus from negative to positive 56 days after vaccination. Seropositivity was defined as an optical density ratio ≥ 1.10, measured using a commercial ELISA. Participants with equivocal serostatus at baseline are counted as non-responders.
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 270 | 265
percentage of participants | 96.7 [93.8 to 98.5] | 95.1 [91.8 to 97.4]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; Difference = 1.6, 95% CI 2-sided [-1.8 to 4.9] — Group 1 - Group 2

8. Secondary Outcome: Seroconversion Rate for Rubella 56 Days Post-vaccination
Description: The seroconversion rate for rubella at 56 days post-vaccination was defined as the percentage of participants with a change in serostatus from negative to positive 56 days after vaccination or a four-fold rise in concentration 56 days after vaccination if seropositive for rubella at baseline. Seropositivity is defined as a post-vaccination concentration of ≥ 10 IU/mL measured using a commercial ELISA.
Time Frame: 56 days after MMR dose 1 vaccination (Day 56)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 285 | 295
percentage of participants | 100.0 [98.7 to 100.0] | 99.7 [98.1 to 100.0]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; Difference = 0.3, 95% CI 2-sided [-0.3 to 1.0] — Group 1 - Group 2

9. Secondary Outcome: Percentage of Participants With Japanese Encephalitis Seropositivity 28 Days Post-vaccination
Description: Japanese encephalitis (JE) immunogenicity was assessed by the percentage of participants with demonstrated seropositivity 28 days after CD-JEV vaccination. Seropositivity was defined as an anti-JE serum neutralizing antibody titer of ≥ 1:10, as measured by JE PRNT-50.
Time Frame: 28 days after CD-JEV vaccination (Day 28 for Group 1 and Day 84 for Group 2)
Population: The JE per-protocol population included participants who fulfilled eligibility criteria, received all study vaccines as assigned, provided valid JE serology results at baseline and 28 days post-vaccination with CD-JEV, did not take any prohibited concomitant medications within 28 days post-vaccination, and did not show JE seropositivity at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 314 | 305
percentage of participants | 72.3 [67.0 to 77.2] | 68.2 [62.6 to 73.4]
Statistical Analysis 1: Comparison: Group 1: MMR and CD-JEV vs Group 2: MMR Then CD-JEV; Test type: Other; Difference = 4.1, 95% CI 2-sided [-3.1 to 11.3]

10. Secondary Outcome: Geometric Mean Titer (GMT) for Serum Neutralizing Antibody Titer to JE Virus at 28 Days Post-vaccination
Description: Anti-JE serum neutralizing antibody titer was measured using JE PRNT-50.
Time Frame: 28 days after CD-JEV vaccination (Day 28 for Group 1 and Day 84 for Group 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Group 1 - MMR and CD-JEV: Participants received one dose of CD-JEV vaccine and one dose of MMR vaccine concurrently at Day 0; Participants received a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
- Group 2 - MMR Then CD-JEV: Participants received one dose of MMR vaccine at Day 0 and one dose of CD-JEV 56 days later. Participants received a second dose of MMR per the routine immunization schedule at Day 84 (12 months of age).
Arm/Group | Group 1 - MMR and CD-JEV | Group 2 - MMR Then CD-JEV
Number analyzed (Participants) | 314 | 305
titer | 24.0 [20.8 to 27.6] | 20.3 [17.8 to 23.1]
Statistical Analysis 1: Comparison: Group 1 - MMR and CD-JEV vs Group 2 - MMR Then CD-JEV; Test type: Other; GMT Ratio = 1.2, 95% CI 2-sided [1.0 to 1.4] — Group 1 / Group 2 ratio obtained using an analysis of covariance (ANCOVA) method with log 10-transformed antibody concentration as dependent variable and treatment group as explanatory variable adjusted for log 10-transformed baseline antibody titer

11. Secondary Outcome: Number of Participants With Immediate Reactions Within 30 Minutes of Each Vaccination
Description: Participants were observed for 30 minutes after each vaccination for immediate reactions. Immediate reactions included both local (injection site) and systemic reactions. MMR vaccine was injected on left upper thigh and CD-JEV was injected on right upper thigh.
  Serious reactions were those meeting one of the following conditions:
  * Death.
  * Life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in a persistent or significant disability or incapacity.
  * Important medical events that, based upon appropriate medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: 30 minutes following each study vaccination
Population: The safety population included all participants who received a study vaccine and had at least one safety measure post-vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: MMR Dose 1 + CD-JEV: Participants in Group 1 received one dose of CD-JEV vaccine and one dose of MMR vaccine concurrently on Day 0.
- Group 2: MMR Dose 1: Participants in Group 2 received one dose of MMR vaccine on Day 0.
- Group 2: CD-JEV: Participants in Group 2 received one dose of CD-JEV on Day 56.
- Group 1: MMR Dose 2: Participants in Group 1 received a second dose of MMR vaccine on Day 84.
- Group 2: MMR Dose 2: Participants in Group 2 received a second dose of MMR vaccine on Day 84.
Arm/Group | Group 1: MMR Dose 1 + CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
Number analyzed (Participants) | 314 | 314 | 309 | 313 | 311
Participants
  Any immediate reaction | 6 | 3 | 5 | 5 | 3
  MMR local reaction: number analyzed (Participants) | 314 | 314 | 0 | 313 | 311
  MMR local reaction | 3 | 2 |  | 3 | 1
  CD-JEV local reaction: number analyzed (Participants) | 314 | 0 | 309 | 0 | 0
  CD-JEV local reaction | 3 |  | 4 |  |
  Systemic | 1 | 1 | 1 | 1 | 2
  Serious reactions | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Solicited Local and Systemic Reactions Within 14 Days of Each Vaccination
Description: Reactogenicity post-vaccination was assessed from 30 minutes through 14 days following vaccination.
  Parents used a structured reactogenicity diary card to record the following solicited (pre-listed) local and system reactions.
  Local reactions (at injection site):
  * Ecchymosis (bruising)
  * Erythema (redness)
  * Edema (swelling)
  * Induration (hardness)
  * Pain/tenderness
  Systemic reactions:
  * Fever
  * Rash
  * Cough
  * Runny nose
  * Change in eating habits
  * Diarrhea
  * Sleepiness
  * Irritability
  * Unusual crying
  * Vomiting
Time Frame: 30 minutes through 14 days following each vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MMR Dose 1 + CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
Number analyzed (Participants) | 314 | 314 | 309 | 313 | 311
Participants
  Any local reactions at MMR injection site: number analyzed (Participants) | 314 | 314 | 0 | 313 | 311
  Any local reactions at MMR injection site | 35 | 31 |  | 12 | 9
  Any local reactions at CD-JEV injection site: number analyzed (Participants) | 314 | 0 | 309 | 0 | 0
  Any local reactions at CD-JEV injection site | 34 |  | 13 |  |
  Any systemic reactions | 224 | 222 | 190 | 168 | 174

13. Secondary Outcome: Number of Participants With Solicited Local Reactions Within 14 Days of Each Vaccination by Maximum Severity
Description: Parents recorded local reactions on a diary card.
  Local ecchymosis, erythema, edema, and induration were graded as follows:
  Grade 1: ≤2.5 cm in diameter.
  Grade 2: >2.5 cm in diameter with 50% of surface area of extremity segment involved.
  Grade 3: ≥50% surface area of extremity segment involved OR ulceration OR secondary infection OR phlebitis OR sterile abscess OR drainage.
  Grade 4: potentially life-threatening (e.g., abscess, exfoliative dermatitis, necrosis involving dermis or deeper tissue).
  Injection site pain/tenderness (pain without touching or tenderness when the area is touched) were graded as follows:
  Grade 1: pain/tenderness causing no or minimal limitation of use of limb. Grade 2: pain/tenderness causing greater than minimal limitation of use of limb.
  Grade 3: pain/tenderness causing inability to perform usual social and functional activities.
  Grade 4: pain/tenderness causing inability to perform basic self-care OR hospitalization indicated.
Time Frame: 30 minutes through 14 days following each vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: MMR Dose 1: Participants in Group 1 received one dose of MMR vaccine injected on the left upper thigh on Day 0.
- Group 1: CD-JEV: Participants in Group 1 received one dose of CD-JEV vaccine injected on the right upper thigh on Day 0.
- Group 2: MMR Dose 1: Participants in Group 2 received one dose of MMR vaccine injected on the left upper thigh on Day 0.
- Group 2: CD-JEV: Participants in Group 2 received one dose of CD-JEV vaccine injected on the left upper thigh on Day 56.
- Group 1: MMR Dose 2: Participants in Group 1 received a 2nd dose of MMR vaccine injected on the left upper thigh on Day 84.
- Group 2: MMR Dose 2: Participants in Group 2 received a 2nd dose of MMR vaccine injected on the left upper thigh on Day 84.
Arm/Group | Group 1: MMR Dose 1 | Group 1: CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
Number analyzed (Participants) | 314 | 314 | 314 | 309 | 313 | 311
Participants
  Ecchymosis: Any | 6 | 6 | 10 | 3 | 0 | 5
  Ecchymosis: Grade 1 | 6 | 6 | 10 | 3 | 0 | 5
  Ecchymosis: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0
  Ecchymosis: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Ecchymosis: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Any | 15 | 13 | 14 | 8 | 5 | 7
  Erythema: Grade 1 | 15 | 12 | 14 | 8 | 5 | 7
  Erythema: Grade 2 | 0 | 1 | 0 | 0 | 0 | 0
  Erythema: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Any | 6 | 3 | 7 | 5 | 0 | 4
  Edema: Grade 1 | 5 | 3 | 7 | 5 | 0 | 4
  Edema: Grade 2 | 1 | 0 | 0 | 0 | 0 | 0
  Edema: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Edema: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Induration: Any | 4 | 7 | 7 | 4 | 0 | 3
  Induration: Grade 1 | 4 | 6 | 7 | 4 | 0 | 3
  Induration: Grade 2 | 0 | 1 | 0 | 0 | 0 | 0
  Induration: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Induration: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Any | 18 | 18 | 19 | 6 | 8 | 5
  Pain/Tenderness: Grade 1 | 17 | 17 | 17 | 5 | 8 | 4
  Pain/Tenderness: Grade 2 | 1 | 1 | 2 | 1 | 0 | 1
  Pain/Tenderness: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Systemic Reactions Within 14 Days of Each Vaccination by Maximum Severity
Description: Parents recorded systemic reactions on a diary card.
  Fever was recorded and graded as follows (axillary temperature):
  Grade 1: 37.5°C to 37.9°C
  Grade 2: 38.0°C to 38.4°C
  Grade 3: 38.5°C to 40.0°C
  Grade 4: >40.0°C
  Rash, cough, runny nose, change in eating habits, diarrhea, sleepiness, irritability, unusual crying, vomiting, and any other unsolicited reaction occurring from 30 minutes through 14 days post vaccination were graded as follows:
  Grade 1: symptoms causing no or minimal interference with usual social and functional activities.
  Grade 2: symptoms causing greater than minimal interference with usual social and functional activities.
  Grade 3: symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated.
  Grade 4: symptoms causing inability to perform basic self-care functions OR medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death.
Time Frame: 30 minutes through 14 days following each vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: MMR Dose 1 + CD-JEV: Participants in Group 1 received one dose of MMR vaccine and one dose of CD-JEV concurrently on Day 0.
- Group 2: CD-JEV: Participants in Group 2 received one dose of CD-JEV vaccine on Day 56.
Arm/Group | Group 1: MMR Dose 1 + CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
Number analyzed (Participants) | 314 | 314 | 309 | 313 | 311
Participants
  Fever: Any | 135 | 119 | 87 | 79 | 84
  Fever: Grade 1 | 52 | 35 | 39 | 31 | 25
  Fever: Grade 2 | 38 | 43 | 21 | 23 | 26
  Fever: Grade 3 | 44 | 40 | 26 | 25 | 32
  Fever: Grade 4 | 1 | 1 | 1 | 0 | 1
  Rash: Any | 27 | 33 | 13 | 19 | 18
  Rash: Grade 1 | 23 | 28 | 12 | 16 | 16
  Rash: Grade 2 | 3 | 4 | 1 | 2 | 2
  Rash: Grade 3 | 0 | 1 | 0 | 0 | 0
  Rash: Grade 4 | 1 | 0 | 0 | 1 | 0
  Cough: Any | 127 | 116 | 118 | 111 | 103
  Cough: Grade 1 | 103 | 92 | 98 | 95 | 90
  Cough: Grade 2 | 20 | 22 | 18 | 16 | 13
  Cough: Grade 3 | 4 | 2 | 2 | 0 | 0
  Cough: Grade 4 | 0 | 0 | 0 | 0 | 0
  Runny nose: Any | 167 | 163 | 143 | 133 | 135
  Runny nose: Grade 1 | 139 | 138 | 128 | 117 | 119
  Runny nose: Grade 2 | 26 | 23 | 14 | 14 | 16
  Runny nose: Grade 3 | 2 | 2 | 1 | 2 | 0
  Runny nose: Grade 4 | 0 | 0 | 0 | 0 | 0
  Change in eating habits: Any | 49 | 32 | 27 | 36 | 27
  Change in eating habits: Grade 1 | 40 | 25 | 23 | 29 | 21
  Change in eating habits: Grade 2 | 9 | 6 | 4 | 6 | 5
  Change in eating habits: Grade 3 | 0 | 1 | 0 | 1 | 1
  Change in eating habits: Grade 4 | 0 | 0 | 0 | 0 | 0
  Diarrhea: Any | 58 | 49 | 29 | 34 | 36
  Diarrhea: Grade 1 | 49 | 45 | 23 | 30 | 25
  Diarrhea: Grade 2 | 7 | 2 | 5 | 1 | 9
  Diarrhea: Grade 3 | 1 | 0 | 1 | 2 | 1
  Diarrhea: Grade 4 | 1 | 2 | 0 | 1 | 1
  Sleepiness: Any | 43 | 32 | 12 | 15 | 16
  Sleepiness: Grade 1 | 39 | 29 | 12 | 15 | 15
  Sleepiness: Grade 2 | 4 | 3 | 0 | 0 | 1
  Sleepiness: Grade 3 | 0 | 0 | 0 | 0 | 0
  Sleepiness: Grade 4 | 0 | 0 | 0 | 0 | 0
  Irritability: Any | 80 | 63 | 36 | 46 | 33
  Irritability: Grade 1 | 63 | 51 | 32 | 40 | 30
  Irritability: Grade 2 | 14 | 10 | 4 | 4 | 2
  Irritability: Grade 3 | 3 | 2 | 0 | 2 | 1
  Irritability: Grade 4 | 0 | 0 | 0 | 0 | 0
  Unusual crying: Any | 54 | 29 | 20 | 29 | 20
  Unusual crying: Grade 1 | 45 | 23 | 17 | 24 | 16
  Unusual crying: Grade 2 | 8 | 5 | 3 | 5 | 3
  Unusual crying: Grade 3 | 1 | 1 | 0 | 0 | 1
  Unusual crying: Grade 4 | 0 | 0 | 0 | 0 | 0
  Vomiting: Any grade | 29 | 26 | 21 | 22 | 31
  Vomiting: Grade 1 | 25 | 18 | 17 | 16 | 20
  Vomiting: Grade 2 | 4 | 8 | 4 | 3 | 9
  Vomiting Grade 3 | 0 | 0 | 0 | 2 | 1
  Vomiting: Grade 4 | 0 | 0 | 0 | 1 | 1

15. Secondary Outcome: Number of Participants With Unsolicited Adverse Events Within 28 Days of Each Vaccination
Description: Each adverse event (AE) was assessed for relationship to vaccine by the study clinician according to the following:
  Definitely Related: An adverse event or unanticipated problem clearly related to the research procedures.
  Possibly Related: There is a reasonable possibility that the adverse event or unanticipated problem, incident, experience, or outcome may have been caused by the procedures involved in the research.
  Not Related: Any adverse event or unanticipated problem clearly not related to study procedures.
  Related adverse events includes events that were assessed as definitely or possibly related.
Time Frame: 28 days following each vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: MMR Dose 1: Participants in Group 2 received one dose of MMR vaccine at Day 0.
Arm/Group | Group 1: MMR Dose 1 + CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
Number analyzed (Participants) | 314 | 314 | 309 | 313 | 311
Participants
  Any adverse event | 207 | 211 | 164 | 110 | 148
  Related adverse events | 35 | 22 | 20 | 22 | 30

16. Secondary Outcome: Number of Participants With Serious Adverse Events Throughout the Study
Description: A serious adverse event (SAE) was defined as an AE that met one of the following:
  * Death
  * Life threatening
  * Required inpatient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability or incapacity
  * Important medical events that, based upon appropriate medical judgment, jeopardized the participant and required medical or surgical intervention to prevent an outcomes listed above
  AEs were assessed for relationship to vaccine by the study clinician according to the following:
  Definitely Related: An AE or unanticipated problem clearly related to the research procedures.
  Possibly Related: There is a reasonable possibility that the AE or unanticipated problem, incident, experience, or outcome may have been caused by the procedures involved in the research.
  Not Related: Any AE or unanticipated problem clearly not related to study procedures.
  Related SAEs includes events that were assessed as definitely or possibly related.
Time Frame: Up to 112 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: MMR and CD-JEV: Participants received one dose of CD-JEV vaccine and one dose of MMR vaccine concurrently on Day 0. Participants received a second dose of MMR per the routine immunization schedule on Day 84 (12 months of age).
- Group 2: MMR Then CD-JEV: Participants received one dose of MMR vaccine on Day 0 and one dose of CD-JEV 56 days later. Participants received a second dose of MMR per the routine immunization schedule on Day 84 (12 months of age).
Arm/Group | Group 1: MMR and CD-JEV | Group 2: MMR Then CD-JEV
Number analyzed (Participants) | 314 | 314
Participants
  Any serious adverse event | 8 | 15
  Related serious adverse event | 0 | 0

ADVERSE EVENTS:
Time Frame: Mortality and serious adverse events were collected through the end of study, up to 112 days. Non-serious adverse events were collected through 28 days after each vaccination.
Arm/Group | Group 1: MMR Dose 1 + CD-JEV | Group 2: MMR Dose 1 | Group 2: CD-JEV | Group 1: MMR Dose 2 | Group 2: MMR Dose 2
All-Cause Mortality (participants affected / at risk) | 0/314 | 0/314 | 0/309 | 0/313 | 0/311
Serious Adverse Events (participants affected / at risk) | 6/314 | 12/314 | 3/309 | 2/313 | 1/311
Other Adverse Events (participants affected / at risk) | 207/314 | 211/314 | 164/309 | 110/313 | 147/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MMR Dose 1 + CD-JEV (N=314) | Group 2: MMR Dose 1 (N=314) | Group 2: CD-JEV (N=309) | Group 1: MMR Dose 2 (N=313) | Group 2: MMR Dose 2 (N=311)
Amoebiasis (Infections and infestations) | 0 | 3 | 0 (0) | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 3 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 2 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: MMR Dose 1 + CD-JEV (N=314) | Group 2: MMR Dose 1 (N=314) | Group 2: CD-JEV (N=309) | Group 1: MMR Dose 2 (N=313) | Group 2: MMR Dose 2 (N=311)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 2 | 5 | 8 | 5
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 4 | 2 | 1 | 2 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 5 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 16 | 24 | 20 | 13 | 15
Bullous impetigo (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 2 | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 4 | 1 | 3 | 1
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 5 | 6 | 1 | 2 | 2
Erythema infectiosum (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 31 | 22 | 19 | 10 | 24
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 6 | 8 | 5 | 1
Herpangina (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Impetigo (Infections and infestations) | 6 | 1 | 4 | 1 | 1
Ludwig angina (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 21 | 19 | 16 | 5 | 13
Oral candidiasis (Infections and infestations) | 0 | 1 | 2 | 0 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 2 | 1 | 3 | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 2 | 3 | 1 | 2 | 2
Pneumonia (Infections and infestations) | 11 | 9 | 6 | 9 | 5
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 31 | 39 | 34 | 17 | 21
Roseola (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 76 | 77 | 54 | 40 | 62
Upper respiratory tract infection bacterial (Infections and infestations) | 6 | 4 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 1 | 3
Varicella (Infections and infestations) | 2 | 4 | 3 | 1 | 0
Viral infection (Infections and infestations) | 24 | 21 | 12 | 8 | 6
Viral rash (Infections and infestations) | 5 | 5 | 0 | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 8 | 9 | 1 | 0 | 0
Wound infection (Infections and infestations) | 6 | 3 | 3 | 3 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Food intolerance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Irritability (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 2 | 2
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT02880865/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02880865/SAP_001.pdf